CLINICAL TRIAL: NCT00694408
Title: A Randomized Pilot Trial of a Steroid-free Immunosuppressant Regimen in Pediatric Liver Transplantation
Brief Title: A Pilot Trial of Pediatric Liver Transplantation Without Steroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to withdrawal from market of Daclizumab
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFPT/OL
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Evidence of Liver Transplantation
Keywords: End stage liver disease; Paediatric liver transplantation; Steroid free immunosuppression
MeSH Terms: conditions — End Stage Liver Disease | interventions — Hydrocortisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid immunosuppressive regimen (Active Comparator): Freedom from rejection and safety in children undergoing paediatric liver transplant using steroid containing immunosuppression regimen post transplant. This group of patients will receive steroids in conjunction with other prescribed immunosuppressive agents. Intervention is use of methyl prednisolone, hydrocortisone, prednisolone as routine post transplant management
  Interventions: Drug: methyl prednisolone, hydrocortisone, prednisolone
- Steroid free immunosuppressive regimen (Active Comparator): Freedom from rejection and safety in children undergoing paediatric liver transplant using steroid free immunosuppression regimen post transplant. The patients in this arm will receive immunosuppression but not steroids to compare with those treated with steroids to measure differences in rejection and safety of a steroid free immunosuppressive regimen. Intervention is omission of methyl prednisolone, hydrocortisone, prednisolone as routine post transplant management. No steroids will be used routinely in this arm
  Interventions: Other: No steroids

INTERVENTIONS:
Drug: methyl prednisolone, hydrocortisone, prednisolone — Will be specific dependant on weight of patients
  Other Names: Methylprednisolone;Hydrocortisone;Prednisolone
  Arms: Steroid immunosuppressive regimen
Other: No steroids — Children undergoing primary liver transplant will receive monoclonal antibodies and tacrolimus as per protocol
  Arms: Steroid free immunosuppressive regimen

SUMMARY:
Objective:

The overall objective is to investigate whether a steroid free immunosuppressive regimen is as safe and effective as a steroid containing regimen following pediatric liver transplantation and whether it promotes tolerance.

DETAILED DESCRIPTION:
3.2 Research question

Is it possible to avoid the use of corticosteroids in pediatric liver transplantation?

3.3 Trial objectives

This will be a pilot study to

i) investigate to what degree a steroid free immunosuppressive regimen is as safe and effective as a steroid containing regimen following pediatric liver transplantation

ii) investigate the effect of a steroid free immunosuppressive regimen on lymphocyte function and donor-specific immune responsiveness following pediatric liver transplantation

iii) investigate the effect of a steroid free immunosuppressive regimen on expression of tissue markers of tolerance following pediatric liver transplantation

It is hoped that this pilot study will be used to develop a definitive multicentre study of a steroid free regimen.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing primary isolated hepatic transplantation.
* Age <=18 years
* Ability to provide informed consent

Exclusion Criteria:

* Children undergoing retransplantation.
* Transplantation for Intestinal failure associated liver disease.
* Multi-organ transplantation.
* Transplantation for autoimmune liver disease.
* Transplantation for extra hepatic malignancy.
* Pre-existing need for oral steroids, or high dose inhaled steroids sufficient to require a steroid warning card.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: The development of histologically proven acute rejection. (within 12 months | 12m

SECONDARY OUTCOMES:
The development of steroid resistant acute rejection 12 months. The expression of tissue and circulating markers of immune tolerance in first year post transplant The incidence of infection in the first year post transplant | 12m

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McKiernan, MRCP FRCPCH, Principal Investigator — Birmingham Children's Hospital
Locations (1):
- Birmingham Children's Hospital, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Sarwal MM, Vidhun JR, Alexander SR, Satterwhite T, Millan M, Salvatierra O Jr. Continued superior outcomes with modification and lengthened follow-up of a steroid-avoidance pilot with extended daclizumab induction in pediatric renal transplantation. Transplantation. 2003 Nov 15;76(9):1331-9. doi: 10.1097/01.TP.0000092950.54184.67. PMID 14627912
- [Background] Vidhun JR, Sarwal MM. Corticosteroid avoidance in pediatric renal transplantation. Pediatr Nephrol. 2005 Mar;20(3):418-26. doi: 10.1007/s00467-004-1786-4. Epub 2005 Feb 3. PMID 15690189
- [Background] Leonard H, Hornung T, Parry G, Dark JH. Pediatric cardiac transplant: results using a steroid-free maintenance regimen. Pediatr Transplant. 2003 Feb;7(1):59-63. doi: 10.1034/j.1399-3046.2003.00014.x. PMID 12581330
- [Background] Walsh PT, Taylor DK, Turka LA. Tregs and transplantation tolerance. J Clin Invest. 2004 Nov;114(10):1398-403. doi: 10.1172/JCI23238. PMID 15545987
- [Background] Yoshizawa A, Ito A, Li Y, Koshiba T, Sakaguchi S, Wood KJ, Tanaka K. The roles of CD25+CD4+ regulatory T cells in operational tolerance after living donor liver transplantation. Transplant Proc. 2005 Jan-Feb;37(1):37-9. doi: 10.1016/j.transproceed.2004.12.259. PMID 15808539
- [Background] Hathaway M, Adams DH. Demonstration that donor-specific nonresponsiveness in human liver allograft recipients is both rare and transient. Transplantation. 2004 Apr 27;77(8):1246-52. doi: 10.1097/01.tp.0000121136.84965.35. PMID 15114093
- [Background] Arora-Gupta N, Davies P, McKiernan P, Kelly DA. The effect of long-term calcineurin inhibitor therapy on renal function in children after liver transplantation. Pediatr Transplant. 2004 Apr;8(2):145-50. doi: 10.1046/j.1399-3046.2003.00132.x. PMID 15049794
- [Background] Evans HM, McKiernan PJ, Kelly DA. Mycophenolate mofetil for renal dysfunction after pediatric liver transplantation. Transplantation. 2005 Jun 15;79(11):1575-80. doi: 10.1097/01.tp.0000163504.29054.3f. PMID 15940048
- [Background] Kelly D, Jara P, Rodeck B, Lykavieris P, Burdelski M, Becker M, Gridelli B, Boillot O, Manzanares J, Reding R. Tacrolimus and steroids versus ciclosporin microemulsion, steroids, and azathioprine in children undergoing liver transplantation: randomised European multicentre trial. Lancet. 2004 Sep 18-24;364(9439):1054-61. doi: 10.1016/S0140-6736(04)17060-8. PMID 15380964
- [Background] Reding R, Gras J, Sokal E, Otte JB, Davies HF. Steroid-free liver transplantation in children. Lancet. 2003 Dec 20;362(9401):2068-70. doi: 10.1016/S0140-6736(03)15104-5. PMID 14697809